CLINICAL TRIAL: NCT03679182
Title: A Pilot Study on Efficacy and Safety of Olanzapine for the Treatment of Nausea and Vomiting in Palliative Cancer Care
Brief Title: Efficacy and Safety of Olanzapine for the Treatment of Nausea and Vomiting in Palliative Cancer Care
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Jarin Chindaprasirt, Assistant professor, Khon Kaen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HE591547
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Nausea; Vomiting; End Stage Cancer
MeSH Terms: conditions — Nausea; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Olanzapine (Experimental): Olanzapine 5 mg at 0, 12, 24 and 36 hours
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine 5 mg Tab at 0, 12, 24, and 36 hours
  Other Names: olanzapine 5 mg Tab

SUMMARY:
Oral olanzapine showed superior antiemetic efficacy to metoclopramide as rescue treatment to control breakthrough emesis induced by chemotherapy. This study aims to evaluate safety and efficacy of olanzapine for nausea and vomiting in advanced cancer patients.

DETAILED DESCRIPTION:
This will be a pilot study; open-label prospective clinical trial. Oral olanzapine 5 mg tablet will be given to patients who fail two standard treatment medications for nausea and vomiting within 30 minutes after the first vomiting episode. Other doses of olanzapine will be given at 12, 24, and 36 hours following the first dose concurrently with standard regimen.

Patients with emesis will be followed up after receiving olanzapine every 12 hour for 48 hours. We will record the frequency of vomiting, nausea, and retching.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years.
2. Diagnosis of advanced malignancy.
3. Failed two standard medications for nausea/vomiting (after 6 hours from last dose).
4. Adequate organ function, including the following:

   1. Hepatic: bilirubin ≤1.5 times the upper limit of normal (x ULN); aspartate aminotransferase (AST), and alanine aminotransferase (ALT) ≤3.0 x ULN (AST, and ALT ≤5 x ULN is acceptable if liver has tumor involvement), alkaline phosphatase (AP) ≤5.0 x ULN.
   2. Renal: calculated creatinine clearance (CrCl) ≥30 mL/min based on the original weight based Cockcroft and Gault formula.
5. Expected life expectancy > 1 month.
6. Patients must be able to read Thai.
7. Patients must sign an informed consent document.

Exclusion Criteria:

1. Patients with history of abdominal radiotherapy.
2. Patients who receive chemotherapy within 1 week.
3. Patients who take fluoxetine.
4. Patients with heart failure or myocardial infarction in the past 6 months.
5. Patients with QTc prolongation from baseline ECG.
6. Known hypersensitivity to olanzapine.
7. Patients who are unwilling to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Emesis control | 48 hours
  Percentage of patients without emesis

CONTACTS AND LOCATIONS:
Overall Officials: Attakorn Raksasataya, MD, Study Director — Khon Kaen University
Locations (1):
- Jarin Chindaprasirt, Khon Kaen, Thailand